CLINICAL TRIAL: NCT03234582
Title: Comparison of Right Ventricular Outflow Tract Gradient Under Anaesthesia With Post-operative Gradient in Patients Undergoing Tetralogy of Fallot Repair
Brief Title: Comparison of RVOT Gradient Under Anaesthesia With Post-operative Gradient in Patients Undergoing TOF Repair
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr. Dheemta Toshkhani, Junior Resident, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: NK/3021/pH/110
Record Dates: First submitted 2017-07-09; First posted 2017-07-31 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Tetralogy of Fallot
MeSH Terms: conditions — Tetralogy of Fallot

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of the study will be to compare intraoperative post TOF repair RVOT gradient under two different anaesthetic depths. Secondary objectives will be to follow up change in RVOT gradient till 1 month post-operatively, observe extubation time, inotropes used post-operatively by vasoactive- inotropic score (VIS), RV functions at discharge from ICU and at 1 month follow- up

DETAILED DESCRIPTION:
After completion of the TOF repair and rewarming to normothermia, all the patients will be assessed by TEE for adequacy of repair and separated from the cardiopulmonary bypass using vasopressors and inotropes. The choice of vasoactive and inotropic agents will be as per the requirement to maintain stable hemodynamics of the patients. Post bypass sevoflurane 1% end tidal concentration (0.5 MAC) will be used in all the patients. RV pressure and gradients across RVOT will be measured directly by placing a 23 gauge needle into the RV and pulmonary artery, and also by TEE using Bernoulli's equation by placing continuous Doppler across tricuspid regurgitation jet and RVOT, as is being routinely done for patients undergoing TOF repair. In addition, velocity time integral (VTI) across left ventricular outflow tract (LVOT) will also be recorded along with other hemodynamic parameters such as HR, SBP, DBP, MAP and SpO2. Subsequently, these measurements will be repeated again after increasing the sevoflurane to 2% end tidal concentration (1 MAC) and allowing the patients to stabilise on this new concentration for 5 minutes while maintaining systemic pressure within a range of 5% of the previous value. Normocarbia (EtCO2 30-35 mmHg) will be maintained during these measurements by adequate minute ventilation.

Following the surgery, all the patients will be shifted to cardio-surgical ICU and will be extubated once they meet the extubation criteria. Post-operative RVOT pressure gradient and RV functions will be assessed by trans-thoracic echocardiography at 2 hrs post extubation, at discharge from ICU and after 1 month of surgery on first follow-up. RV functions on echocardiography will be assessed using TAPSE (Tricuspid annular plane systolic excursion) and fractional RV area change during systole. The duration of post-operative mechanical ventilation, vasoactive inotropic score (VIS), PaO2/FiO2 ratio till discharge from ICU and any morbidity or adverse outcome during hospital stay will be noted.

ELIGIBILITY:
Inclusion Criteria:

* All the children between 6 months to 16 years of age undergoing TOF repair will be included in the study.

Exclusion Criteria:

* TOF patients with pulmonary atresia, atrioventricular canal defects and where consent is refused will be excluded from the study.

Ages: 6 Months to 16 Years | Sex: All
Age Groups: Child
Study Population: All the children between 6 months to 16 years of age undergoing TOF repair will be included in the study.TOF patients with pulmonary atresia, atrioventricular canal defects and where consent is refused will be excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-08-01 (Estimated); Study Completion 2018-08-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of right ventricular outflow tract gradient under anaesthesia with post-operative gradient in patients undergoing tetralogy of Fallot repair | 15 minutes
  The primary objective of the study will be to compare intra-operative post TOF repair RVOT gradient under two different anaesthetic depths

SECONDARY OUTCOMES:
Comparison of change in right ventricular outflow tract gradient post-operatively in patients undergoing tetralogy of Fallot repair | 1 month
  To follow up change in RVOT gradient till 1 month post-operatively, observe extubation time, inotropes use post-operatively by vasoactive-inotropic score (VIS), RV functions at discharge from ICU and at 1 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Dheemta Toshkhani, MD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Nandita Kakkar, Chandigarh, India

REFERENCES:
- [Derived] Toshkhani D, Arya VK, Kajal K, Thingnam SKS, Rana SS. Comparison of right ventricular outflow tract gradient under anesthesia with post-operative gradient in patients undergoing tetralogy of Fallot repair. Ann Pediatr Cardiol. 2021 Jan-Mar;14(1):18-25. doi: 10.4103/apc.APC_147_19. Epub 2020 Oct 19. PMID 33679057